CLINICAL TRIAL: NCT02277054
Title: A Clinical Trial to Evaluate the Safety and Effectiveness of the Collagen-phosphorylcholine Corneal Substitutes in Patients Requiring Lamellar Keratoplasty
Brief Title: Safety and Effectiveness of Collagen-phosphorylcholine Bioengineered Cornea in Patients Requiring Lamellar Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03/2013
Record Dates: First submitted 2014-10-26; First posted 2014-10-28 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Corneal Ulcer; Leukoma
MeSH Terms: conditions — Corneal Ulcer; Corneal Opacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collagen-MPC cornea substitute (Experimental): Collagen-phosphorylcholine (collagen-MPC) cornea substitute transplantation using anterior lamellar keratoplasty technique.
  Interventions: Device: Collagen-MPC cornea

INTERVENTIONS:
Device: Collagen-MPC cornea — Patients will undergo surgery using conventional anterior lamellar keratoplasty technique: diseased cornea will be trephined to approximately 50-90% of corneal thickness (depending on corneal ulcer or scar depth) and then a lamellar dissection will be created. Trephine diameter will depend on ulcer or leukoma maximal size. Alternatively a femtosecond laser may be used to create the dissection. A collagen-phosphorylcholine cornea 250-500 microns thick and equal or 0.25 mm larger diameter is placed and sutured. The sutures are superimposed and the implant and the sutures covered with a bandage contact lens. The sutures and bandage lens will be removed later after the initial healing period of 4 weeks or as determined by physician depending on the implant epithelial coverage.

SUMMARY:
In this study the safety and effectiveness of biosynthetic cornea, comprising interpenetrating networks of recombinant human collagen and phosphorylcholine, will be tested in patients with severe corneal pathology (corneal ulcers or corneal opacification from corneal injury, burn or infection) - diseases, where human donor cornea transplantation (the only widely accepted treatment) carries a high risk of rejection.

DETAILED DESCRIPTION:
Collagen-phosphorylcholine corneal substitute will be implanted in patient's corneas with severe pathology (corneal ulcer, corneal leukoma after burn, trauma or infection) using anterior lamellar keratoplasty technique, i.e. when patient's diseased cornea is removed it will be substituted with proposed transparent implant. Usually these patients are grafted with human donor cornea, but the latter frequently fails due to graft-versus-host problems. We will test the safety (incidence of adverse events, biocompatability) and the effectiveness (ability to promote healing and increase vision) of developed biosynthetic corneas in 10 patients with corneal pathology, where human donor cornea carries a high risk of rejection. The patients will be follow-uped for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign and be given a copy of the written Informed Consent form.
2. Subjects with best corrected distance visual acuity 20/200 or worse as a result of corneal ulcer or corneal scar due to burn, injury or infection in the operative eye.
3. Subjects must be willing and able to return for scheduled follow-up examinations for 12 months after surgery.

Exclusion Criteria:

1. Subjects with severe or life-threatening systemic disease.
2. Subjects with uncontrolled hypertension.
3. Subjects with uncontrolled diabetes or insulin-dependent diabetes.
4. Subjects with glaucoma in either eye.
5. Subjects with marked microphthalmos or aniridia in either eye.
6. Subjects with any other serious ocular pathology, serious ocular complications at the time of corneal transplant underlying serious medical conditions, based on the investigator's medical judgment.
7. Subjects which are or lactating or who plan to become pregnant over the course of the clinical investigation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Pasyechnikova, MD, PhD, DSc, Study Director — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (1):
- The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu W, Deng C, McLaughlin CR, Fagerholm P, Lagali NS, Heyne B, Scaiano JC, Watsky MA, Kato Y, Munger R, Shinozaki N, Li F, Griffith M. Collagen-phosphorylcholine interpenetrating network hydrogels as corneal substitutes. Biomaterials. 2009 Mar;30(8):1551-9. doi: 10.1016/j.biomaterials.2008.11.022. Epub 2008 Dec 20. PMID 19097643
- [Result] Hackett JM, Lagali N, Merrett K, Edelhauser H, Sun Y, Gan L, Griffith M, Fagerholm P. Biosynthetic corneal implants for replacement of pathologic corneal tissue: performance in a controlled rabbit alkali burn model. Invest Ophthalmol Vis Sci. 2011 Feb 3;52(2):651-7. doi: 10.1167/iovs.10-5224. PMID 20847116

RESULTS

PARTICIPANT FLOW:
Groups:
- RHCIII-MPC Cornea Substitute: Recombinant human collagen type III -methylphosphorylcholine (RHCIII-MPC) cornea substitute transplantation using anterior lamellar keratoplasty technique.
  Patients underwent surgery using conventional anterior lamellar keratoplasty technique: diseased cornea was trephined to approximately 50-90% of corneal thickness (depending on corneal ulcer or scar depth) and then a lamellar dissection was created. Trephine diameter depended on ulcer or leukoma maximal size. A RHCIII-MPC cornea 350 microns thick and equal or 0.25 mm larger diameter was placed and sutured. The sutures were superimposed and the implant and the sutures covered with a bandage contact lens. The sutures and bandage lens were removed later after the initial healing period of 4 weeks or as determined by physician depending on the implant epithelial coverage.
Period: Overall Study
Arm/Group | RHCIII-MPC Cornea Substitute
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- RHCIII-MPC Cornea Substitute: Recombinant human collagen type III -methylphosphorylcholine (RHCIII-MPC) cornea substitute transplantation using anterior lamellar keratoplasty technique.
  Patients underwent surgery using conventional anterior lamellar keratoplasty technique: diseased cornea was trephined to approximately 50-90% of corneal thickness (depending on corneal ulcer or scar depth) and then a lamellar dissection was created. Trephine diameter depended on ulcer or leukoma maximal size. A RHCIII-MPC cornea 250-500 microns thick and equal or 0.25 mm larger diameter was placed and sutured. The sutures are superimposed and the implant and the sutures covered with a bandage contact lens. The sutures and bandage lens were removed later after the initial healing period of 4 weeks or as determined by physician depending on the implant epithelial coverage.
Arm/Group | RHCIII-MPC Cornea Substitute
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ukraine | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Implant safety and tolerability will be measured by absence/presence of its lysis as well as by degree of eye inflammation based on conjunctival injection, perifocal corneal haze, aqueous humor transparency, increased intraocular pressure and self reported postoperative pain. Each item is scored 0-4: 0 = no symptom, 4 = severe symptom.
Time Frame: 12 months
Measure: Number; unit: events
Groups:
- RHCIII-MPC Cornea Substitute: Recombinant human collagen type III-methylphosphorylcholine (RHCIII-MPC) cornea substitute transplantation using anterior lamellar keratoplasty technique.
  Patients underwent surgery using conventional anterior lamellar keratoplasty technique: diseased cornea was trephined to approximately 50-90% of corneal thickness (depending on corneal ulcer or scar depth) and then a lamellar dissection was created. Trephine diameter depended on ulcer or leukoma maximal size. A RHCIII-MPC cornea 350 microns thick and equal or 0.25 mm larger diameter was placed and sutured. The sutures were superimposed and the implant and the sutures covered with a bandage contact lens. The sutures and bandage lens were removed later after the initial healing period of 4 weeks or as determined by physician depending on the implant epithelial coverage.
Arm/Group | RHCIII-MPC Cornea Substitute
Number analyzed (Participants) | 5
events | 0

2. Secondary Outcome: Number of Participants With Healed Cornea at 12 Months
Description: Cornea is considered to have healed up when there is no defect of corneal epithelium, which is confirmed by fluorescein staining of corneal surface
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RHCIII-MPC Cornea Substitute
Number analyzed (Participants) | 5
Participants | 5

3. Secondary Outcome: Number of Participants With Improved Visual Acuity at 12 Months
Description: Improvement of 1 or more lines in Corrected Distance Visual Acuity in comparison to preoperative visual acuity
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RHCIII-MPC Cornea Substitute
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Arm/Group | RHCIII-MPC Cornea Substitute
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes